CLINICAL TRIAL: NCT01110317
Title: Open-Label, Parallel, Randomized, Multiple-Dose Pharmacokinetic Study of Paliperidone After Intramuscular Injection of Paliperidone Palmitate in the Deltoid or Gluteal Muscle in Subjects With Schizophrenia
Brief Title: A Study of Paliperidone Blood Concentrations in Patients With Schizophrenia After Administration of Paliperidone Palmitate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Associate Director, Clinical Pharmacoloy, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002362; R092670PSY1001
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Paliperidone palmitate; R092670PSY1001; Pharmacokinetics; Risperdal (CONSTA); Risperidone, Paliperidone
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

ARMS (1):
- 001 (Experimental): paliperidone palmitate 100 mg Patients will receive a single paliperidone palmitate 100 mg equivalent injection in the gluteal or deltoid muscle on Day 1 8 36 and 64.
  Interventions: Drug: paliperidone palmitate 100 mg

INTERVENTIONS:
Drug: paliperidone palmitate 100 mg — Patients will receive a single paliperidone palmitate 100 mg equivalent injection in the gluteal or deltoid muscle on Day 1, 8, 36, and 64.

SUMMARY:
The purpose of this study is to evaluate the concentration of paliperidone in the blood after intramuscular injection in upper arm (deltoid muscle) or in the buttock (gluteal muscle) in patients with schizophrenia.

DETAILED DESCRIPTION:
This is a an open-label (all patients will know the name of the study drug that they are receiving), randomized (patients will selected by "chance" or like "flipping a coin" to administration of study drug by intramuscular [i.m.] injection into the gluteal [buttocks] or deltoid [upper arm] muscle of the body) study in patients with schizophrenia. A minimum of 40 patients (20 patients per group [1 group of patients to be administered study drug by injection in the gluteal muscle and 1 group of patients to be administered study drug by injection in the deltoid muscle]) will participate in this study, including at least 4 women in each group. The study will consist of a screening period that will occur within 21 days before the first study drug administration, an open-label treatment period during which patients will receive a total of 4 injections of study drug (paliperidone palmitate) either in the deltoid or gluteal muscle, and an end-of-study visit where final study evaluations will be performed. At the screening visit, if a patient has been treated with an antipsychotic medication before study entry, the medication may be continued during the study except for medications specified in the exclusion criteria for the study. If patients have not been previously treated with 1 of the following antipsychotic drugs: risperidone, paliperidone, or paliperidone palmitate, they will undergo a 4-day evaluation period where they will be given a 3 mg/day dose of an extended release (ER) formulation of paliperidone to evaluate their ability to tolerate study drug. Patients who meet all entry criteria for the study will be randomly assigned to 1 of 2 treatment groups in which they will receive 100 mg equivalent of paliperidone palmitate by i.m. injection in either the gluteal muscle or the deltoid muscle. Blood samples for pharmacokinetics (ie, to test the concentration of study drug in the blood) will be collected at specified times before and after each dose of study drug. A single blood sample may also be collected at any time during screening or before the first day of i.m. administration of study drug for patients who agree to participate in an optional part of the study called a pharmacogenomic evaluation which is an evaluation where genetic information obtained from the patient's blood is used to predict whether or not study drug will help make the patient well. During the study, the patient's psychiatric symptoms, severity of symptoms, and injection site reactions will be evaluated. The primary outcome measure in the study will be the determination of the concentration of paliperidone in the patient's blood before study drug administration at protocol-specified time points during the study. The patient's safety will be monitored throughout the study by performing physical examinations, vital signs measurements, clinical laboratory tests, electrocardiograms (ECGs), monitoring of extrapyramidal symptoms (ie, symptoms that can be associated with taking antipsychotic medications), injection site evaluations, and recording of adverse events (side effects). Each patient will receive a total of 4 paliperidone palmitate 100 mg equivalent injections in the gluteal or deltoid muscle on Day 1, 8, 36, and 64.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) for more than 1 year that is clinically stable with no change in current antipsychotic medications for 3 months prior to screening
* Have a total Positive and Negative Syndrome Scale for Schizophrenia (PANSS) score of 70 or less, a score of no more than 16 points on the sum of the following 4 items of the PANSS: conceptual disorganization, suspiciousness/persecution, hallucinatory behavior, and unusual thought content, and scores not greater than 5 on any of the individual items of the PANSS
* Be otherwise healthy confirmed by prestudy physical examination, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory tests
* Sign an informed consent document indicating an understanding of the purpose and procedures required for the study and a willingness to participate in the study

Exclusion Criteria:

* Have a DSM-IV diagnosis of alcohol or substance dependence, with the exception of nicotine or caffeine dependence, within 12 months prior to screening
* Be involuntarily-hospitalized or plan to undergo surgery/procedures during the course of the study
* Take the following prohibited medications: oral risperidone within 2 weeks of randomization, oral paliperidone within 2 weeks of randomization with the exception of the tolerability testing period, clozapine therapy within 6 weeks of randomization, use of ziprasidone and thioridazine within 1 week prior to randomization, risperidone within 100 days of screening, a paliperidone palmitate long-acting preparation within 10 months of randomization, long-acting formulations of other neuroleptic drugs within 1 treatment cycle before screening, barbiturates within 14 days prior to randomization, any anticonvulsant medications within 14 days prior to randomization, or use of irbesartan within 1 week prior to randomization
* Have a history of an allergic reaction to risperidone, paliperidone, or any of their excipients, or have a known hypersensitivity to risperidone or paliperidone
* Have current thoughts of suicide (suicidal ideation) or violent tendencies at the time of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-07; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Determination of the concentration of paliperidone in blood samples obtained from patients. | Predose at specified time points (Days 18, 20, 22, 29, 46, 50, 85, 92, 99, 106, 120, 134, 148, 162, and 176) during the study through Day 176 or the time of early withdrawal from the study.

SECONDARY OUTCOMES:
The safety of paliperidone palmitate i.m. injections in patients will be evaluated by injection site evaluations, clinical laboratory tests, vital signs measurements, and physical examinations. | From time of screening (Visit 1) through the end of study (Visit 33 [Day 176]) or at the time of early withdrawal from the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Rossenu S, Cleton A, Hough D, Crauwels H, Vandebosch A, Berwaerts J, Eerdekens M, Herben V, De Meulder M, Remmerie B, Francetic I. Pharmacokinetic profile after multiple deltoid or gluteal intramuscular injections of paliperidone palmitate in patients with schizophrenia. Clin Pharmacol Drug Dev. 2015 Jul;4(4):270-8. doi: 10.1002/cpdd.144. Epub 2014 Aug 28. PMID 27136907